CLINICAL TRIAL: NCT06936397
Title: A Randomized Controlled EEG-GSR Study on the Effects of Cognitive Remediation Therapy on Neurophysiological and Emotional Regulation Markers in Schizophrenia
Brief Title: Cognitive Remediation Therapy for Schizophrenia: Effects on EEG and Emotional Regulation
Acronym: CRT-SCHZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beykoz University (Other)
Collaborators: Uskudar University (Other); Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Eda Yilmazer, Principle investigator, Beykoz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRT-SCHZ-IST-2025
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia Disorders; Cognitive Dysfunction; Emotion Regulation Disorders
Keywords: Cognitive Remediation Therapy; Schizophrenia; EEG; GSR; Emotion Regulation; Executive Function; P300; Mismatch Negativity; Neurophysiological Biomarkers; Psychophysiology
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Parallel assignment: Schizophrenia participants will be randomized into two groups (CRT intervention vs. waitlist control). Healthy controls will not receive an intervention but will serve as a normative reference group for baseline EEG and GSR measures.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT Group (Experimental): Participants with schizophrenia assigned to receive 12 sessions of Cognitive Remediation Therapy (CRT) over 12 weeks. Each session lasts approximately 60 minutes and targets cognitive domains including attention, working memory, executive function, and emotion regulation.
  Interventions: Behavioral: Cognitive Remediation Therapy
- Waitlist Control (No Intervention): Participants with schizophrenia assigned to a waitlist control group. They will not receive any therapy during the 12-week period but will undergo baseline and post-assessments similar to the CRT group.

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — CRT is a structured behavioral intervention consisting of weekly 60-minute sessions for 12 weeks. The therapy includes tasks to enhance cognitive skills such as attention, memory, executive function, and emotional regulation using computer-based training and therapist-guided exercises.
  Arms: CRT Group

SUMMARY:
This study aims to determine whether Cognitive Remediation Therapy (CRT) can improve attention, memory, and emotional regulation in people with schizophrenia. CRT is a structured program that includes exercises to strengthen cognitive skills such as problem-solving, working memory, and emotion regulation.

The study will recruit 60 participants: 30 individuals with schizophrenia and 30 healthy individuals of similar age and gender. Those with schizophrenia will be randomly assigned to either receive CRT or be placed on a waitlist without therapy. All participants will undergo non-invasive brain activity (EEG) and emotional response (GSR) recordings before and after the therapy.

The study's main question is: Does participating in a 12-week CRT program improve brain-based markers of attention and emotional regulation in people with schizophrenia?

Additional tests, such as memory and emotion recognition tasks and self-report questionnaires, will help assess changes in thinking skills and emotional well-being. The study may help better understand how CRT affects both brain function and quality of life in schizophrenia.

DETAILED DESCRIPTION:
This is a randomized controlled trial examining the effects of Cognitive Remediation Therapy (CRT) on neurophysiological and behavioral outcomes in schizophrenia. The primary goal is to assess whether CRT improves attentional control, sensory processing, executive function, and emotional regulation as measured by EEG and GSR.

Sixty participants will be enrolled: 30 individuals diagnosed with schizophrenia (DSM-5 criteria) and 30 healthy controls matched by age and gender. The schizophrenia group will be randomized into a CRT intervention arm and a waitlist control group. Healthy controls will not undergo CRT but will participate in baseline neurophysiological assessments to establish normative EEG and GSR values.

CRT will consist of 12 weekly sessions (approximately 60 minutes each), targeting cognitive domains such as working memory, attention, executive function, and emotion regulation using structured exercises and computer-based tasks.

EEG recordings will include P300 (oddball paradigm), mismatch negativity (MMN), and frontal theta power (cognitive control tasks). GSR will assess baseline skin conductance and reactivity to negative emotional stimuli. Behavioral tasks include the Stroop task, digit span, and facial emotion recognition.

Psychometric instruments include the Turkish-validated versions of:

* Difficulties in Emotion Regulation Scale (DERS)
* Brief Assessment of Cognition in Schizophrenia (BACS)
* Schizophrenia Quality of Life Scale (SQLS)

Primary outcomes will be assessed via pre- and post-test comparisons. Statistical methods include repeated-measures ANOVA, mixed-effects modeling, and regression analyses linking physiological changes to cognitive and emotional performance.

The study is ethically approved and aligns with international standards for human research.

ELIGIBILITY:
Inclusion Criteria (Schizophrenia Group):

* Diagnosed with schizophrenia according to DSM-5 criteria
* Age between 18 and 55 years
* Clinically stable (no hospitalization or medication change within 1 month)
* Minimum primary school education
* Able to provide informed consent
* Right-handed (for EEG protocol consistency)

Inclusion Criteria (Healthy Control Group):

* No history of psychiatric or neurological disorders
* Age- and gender-matched to schizophrenia group
* No current medication affecting CNS
* Able to provide informed consent
* Right-handed

Exclusion Criteria (Both Groups):

* Current or past substance use disorder (within the past year)
* Comorbid neurological illness (e.g., epilepsy, traumatic brain injury)
* Current use of benzodiazepines or medications that significantly affect cognitive function
* Intellectual disability or MoCA score < 20
* Visual or hearing impairments that could interfere with task performance
* Participation in a psychological intervention in the last 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in P300 Amplitude Measured via EEG at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  P300 amplitude will be recorded during an auditory oddball task using EEG. Increased P300 amplitude after the 12-week CRT intervention is interpreted as an improvement in attentional processing and cognitive engagement. P300 is a continuous electrophysiological variable typically ranging from 0 to 15 microvolts; higher values post-intervention suggest enhanced neurocognitive performance.

SECONDARY OUTCOMES:
Change from Baseline in Mismatch Negativity (MMN) Amplitude Measured via EEG at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  MMN amplitude will be measured during an auditory passive oddball paradigm to assess sensory discrimination and predictive coding. MMN is an event-related potential, with amplitudes typically ranging from 0 to -10 µV. Increased MMN amplitude post-intervention indicates improved auditory processing.
Change from Baseline in Frontal Midline Theta Power During Cognitive Tasks at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  Frontal theta power (4-8 Hz) will be extracted from EEG recordings during cognitive tasks such as the Stroop and n-back. Increases in theta power are associated with enhanced working memory and executive control.
Change from Baseline in Skin Conductance Response (SCR) to Emotional Stimuli at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  GSR responses to emotionally negative images will be measured. A decrease in SCR amplitude reflects reduced emotional hyperreactivity and improved autonomic regulation.
Change from Baseline in Difficulties in Emotion Regulation Scale (DERS) Total Score at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  Self-reported emotion regulation difficulties will be assessed using the Turkish-validated DERS. Scores range from 36 to 180, with higher scores indicating more severe regulation difficulties. A decrease in score post-intervention reflects improved regulation.
Change from Baseline in Brief Assessment of Cognition in Schizophrenia (BACS) Total Score at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  BACS assesses domains such as verbal memory, attention, working memory, and executive function. Higher scores post-intervention indicate improved cognitive performance.
Change from Baseline in Schizophrenia Quality of Life Scale (SQLS) Total Score at 12 Weeks | Baseline and 12 Weeks Post-Intervention
  The SQLS measures subjective quality of life in schizophrenia. Lower total scores after CRT indicate improvements in psychological and social well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Gökben Hızlı Sayar, Professor, Study Chair — Üsküdar University; Selami Varol Ülker, Phd, Study Director — Üsküdar University; Metin Çınaroğlu, Phd, Principal Investigator — İstanbul Nişantaşı University
Locations (1):
- Beykoz University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes (e.g., EEG, GSR, and psychometric scores) will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available beginning 6 months after publication and for up to 5 years.
Access Criteria: Researchers may request access by contacting the Principal Investigator.